CLINICAL TRIAL: NCT00414271
Title: A Phase II Study of Neo-adjuvant Chemotherapy in Locally Advanced Gastric Cancer
Brief Title: Neo-adjuvant Chemotherapy in Locally Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS 0420; NA_00044000 (Other: JHM IRB)
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-05

CONDITIONS: Stage T3-4NxM0 Gastric Cancer
Keywords: gastric cancer, neo-adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Docetaxel and Capecitabine in gastric cancer (Experimental): Intravenous docetaxel 60 mg/m2 on day 1 and oral capecitabine 900 mg/m2 two times per day from day 1 to day 14 every 3 weeks for 2 cycles.
  Interventions: Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 60 mg/m2 IV on day 1
Drug: Capecitabine — Capecitabine 900 mg/m2 PO two times per day from day 1 to day 14 every 3 weeks for 2 cycles.

SUMMARY:
Thymidylate Synthase (TS) is a key enzyme in the synthesis of DNA and the target enzyme inhibited by 5-fluorouracil (5-FU). TS level in the tumour cells has been reported as predictive to response to 5-FU and a prognostic factor in colorectal and gastric cancer patients. We plan to study TS by immunohistochemistry (IHC) in the paraffin blocks of tumour tissue.

A combined comparative genomic hybridization (CGH) and expression microarray analysis of gastric cancer specimens before and after neoadjuvant chemotherapy. CGH will be performed using standard technique routinely done in Dr Patrick Tan's laboratory at the National Cancer Centre, which determines the gain or loss of DNA copies of each chromosome. Total RNA will be extracted from at least one biopsy sample which contains at least 50% cancer cells by homogenization of the tumour tissue and tri-sol method. 5 ug of RNA were amplified and hybridized with the C-DNA microarrays of 18K targets.

Primary Objective 1. Feasibility and safety of pre-operative chemotherapy in locally advanced gastric cancer.

Secondary Objective

1. Complete clinical and pathological response rates to pre-operative chemotherapy in locally advanced gastric cancer
2. Complete resection rate.
3. Time to recurrence, disease free and overall survival
4. Correlation of clinical outcome with (Runt-related transcription factor) RUNX-3 methylation status and Thymidylate synthetase in the tumor tissue.
5. Correlation of CGH and gene expression profile and their changes after chemotherapy with clinical outcome.

   Patients may be included in the study only if they meet all of the following criteria:

   Age at least 18 years. Histologic or cytologic diagnosis of adenocarcinoma of stomach or gastric cardia (Siewert Classification Type III) Preoperative Stage T3-4NxM0 by endoscopic ultrasound, CT of the abdomen/pelvis and laparoscopy. (CT of the chest if it is a cardia lesion).

   Absence of malignant cells in peritoneal lavage fluid during laparoscopic examination.

   Patients must not have received any prior chemotherapy or hormonal therapy for the treatment of gastric cancer.

   Karnofsky performance status of 70 or higher. Estimated life expectancy of at least 12 weeks.

   Adequate organ function including the following:

   - Bone marrow: White blood cells (WBC) at least 3.5 x 109/L Absolute neutrophil (segmented and bands) count (ANC) at least 1.5 x 109/L Platelets at least 100 x 109/L Haemoglobin at least 9g/dL

   - Hepatic: Bilirubin within upper limit of normal (ULN), Aspartate transaminase (ALT) or Alanine transaminase (AST) not more than 2.5x ULN Alkaline phosphatase not more than 2.5x ULN.

   - Renal: creatinine not more than 1.5x ULN Signed informed consent by patient or legal representative. Patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

   The study plans to recruit 30 patients in 12-18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal 18 years.
* Histologic or cytologic diagnosis of adenocarcinoma of stomach or gastric cardia (Siewert Classification Type III)
* Preoperative Stage T3-4NxM0 by endoscopic ultrasound, CT of the abdomen/pelvis and laparoscopy. (CT of the chest if it is a cardia lesion).
* Absence of malignant cells in peritoneal lavage fluid during laparoscopic examination.
* Patients must not have received any prior chemotherapy or hormonal therapy for the treatment of gastric cancer.
* Karnofsky performance status of 70 or higher.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:
* Bone marrow:

  * White blood cells (WBC) greater than or equal 3.5 x 109/L
  * Absolute neutrophil (segmented and bands) count (ANC) greater than or equal 1.5 x 109/L
  * Platelets greater than or equal 100 x 109/L
  * Haemoglobin greater than or equal 9g/dL
* Hepatic:

  * Bilirubin within upper limit of normal (ULN),
  * ALT or AST less than or equal 2.5x ULN
  * Alkaline phosphatase less than or equal 2.5x ULN.
* Renal:

  * creatinine less than or equal 1.5x ULN
* Signed informed consent by patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Prior treatment for locally advanced or metastatic gastric cancer. Any metastatic disease will render patient ineligible according to American Joint Committee on Cancer (AJCC) staging manual. (See appendix 11.4).
* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other cancer therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast-feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Poorly controlled diabetes mellitus with fasting blood sugar > 18 mmol/L(mM).
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* History of significant neurological or mental disorder, including seizures or dementia.
* History of hypersensitivity to drugs formulated in Tween 80, the vehicle used for commercial docetaxel formulations.
* History of hypersensitivity to 5-fluorouracil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chang, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Singapore International Medical Center, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang AY, Foo KF, Koo WH, Ong S, So J, Tan D, Lim KH. Phase II study of neo-adjuvant chemotherapy for locally advanced gastric cancer. BMJ Open Gastroenterol. 2016 Aug 23;3(1):e000095. doi: 10.1136/bmjgast-2016-000095. eCollection 2016. PMID 27648294
- See also: Related Info — https://bmjopengastro.bmj.com/content/3/1/e000095

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Docetaxel and Capecitabine in Gastric Cancer
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: >= 18 years old
Arm/Group | Docetaxel and Capecitabine in Gastric Cancer
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 18
locally advanced gastric cancer [Count of Participants; unit: Participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathological Response
Description: Number of participants who completed neoadjuvant chemotherapy and underwent repeat CT and endoscopic ultrasound (EUS) with pathological complete response (pCR), partial response in the primary tumor, stable disease or progressive disease as defined by EUS criteria.
Time Frame: up to 5 years
Population: Only 15 of the participants who completed neoadjuvant chemotherapy and underwent repeat CT and EUS had measurable tumors by both imaging methods.
Measure: Count of Participants; unit: Participants
Groups:
- Open Label, Single Arm: Capecitabine, docetaxol
Arm/Group | Open Label, Single Arm
Number analyzed (Participants) | 15
Participants
  pathological complete response (pCR) | 0
  partial response | 4
  stable disease | 8
  progressive disease | 3

2. Secondary Outcome: Overall Survival
Description: Median number of months participants alive at the time of observation. Calculated using Kaplan-Meier method.
Time Frame: up to 8 years
Population: 1 participant was lost to follow-up after progression from neoadjuvant chemotherapy.
Measure: Median (Full Range); unit: months
Arm/Group | Open Label, Single Arm
Number analyzed (Participants) | 17
months | 17.1 [7.4 to 84.7]

3. Secondary Outcome: Progression-free Survival as Measured by Number of Participants Without Disease Progression.
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label, Single Arm
Number analyzed (Participants) | 18
Participants | 3

4. Secondary Outcome: Feasibility and Safety of Pre-operative Chemotherapy in Locally Advanced Gastric Cancer as Assessed by Number of Participants Who Experienced Adverse Events Grade 3 or Higher as Defined by CTCAE.
Description: Number of participants who experience Grade 3/4 neutropenia, Grade 3 nausea or Grade 3 diarrhea.
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label, Single Arm
Number analyzed (Participants) | 18
Participants
  Grade 3/4 neutropenia | 10
  Grade 3 nausea | 1
  Grade 3 diarrhea | 2

5. Secondary Outcome: Correlation of CGH and Gene Expression Profile and Their Changes After Chemotherapy With the Same Clinical Outcomes
Description: Initially, we also planned to study the thymidylate synthetase expression, methylation of RUNX-3 gene[24] and comprehensive genomic hybridization[25] before and after chemotherapy to look for biomarkers of response and prognostic indication. But due to the lack of pCR and the small number of patients enrolled, we stopped the correlative studies.
Time Frame: up to 5 years
Population: Data was not collected to assess this outcome measure.
Arm/Group | Open Label, Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Open Label, Single Arm
All-Cause Mortality (participants affected / at risk) | 11/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label, Single Arm (N=18)
Myocardial infarction (Cardiac disorders) | 1 (1) — One patient developed a myocardial infarction after the first cycle of chemotherapy and was taken off protocol.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label, Single Arm (N=18)
Anemia (Blood and lymphatic system disorders) | 2 (2) — Grade 1
Anemia (Blood and lymphatic system disorders) | 2 (2) — Grade 3
Constipation (Gastrointestinal disorders) | 4 (4) — Grade 1
constipation (Gastrointestinal disorders) | 1 (1) — Grade 2
Diarrhoea (Gastrointestinal disorders) | 3 (3) — Grade 1
Diarrhoea (Gastrointestinal disorders) | 4 (4) — Grade 2
Diarrhoea (Gastrointestinal disorders) | 2 (2) — Grade 3
Nausea (Gastrointestinal disorders) | 2 (2) — Grade 1
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 3
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 2
Neutropenia (Blood and lymphatic system disorders) | 4 (4) — Grade 3
Neutropenia (Blood and lymphatic system disorders) | 6 (6) — Grade 4
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) — Grade 1
Fatigue (General disorders) | 2 (2) — Grade1
Myalgia (General disorders) | 3 (3) — Grade 1
Insomnia (General disorders) | 1 (1) — Grade 2
Insomnia (General disorders) | 2 (2) — Grade 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No